CLINICAL TRIAL: NCT05625204
Title: High Intensity Interval Training (HIIT) to Reduce Frailty and Enhance Resilience in Older Veterans
Acronym: HIIT@Home
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E3813-R; RX003813-01A2 (Other Grant/Funding Number: Veterans Affairs)
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Frailty
Keywords: aging; frailty; veteran; functional capacity; resilience; cognition; sleep
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Center based attention control (Experimental): Center based attention control
  Interventions: Behavioral: Center based attention (stretching only) control
- Center based HIIT (Experimental): Center based HIIT
  Interventions: Behavioral: Center based HIIT
- Home based HIIT (Experimental): Home based HIIT
  Interventions: Behavioral: Home based HIIT

INTERVENTIONS:
Behavioral: Center based attention (stretching only) control — Center based attention (stretching only) control
  Arms: Center based attention control
Behavioral: Center based HIIT — Center based HIIT
  Arms: Center based HIIT
Behavioral: Home based HIIT — Home based HIIT
  Arms: Home based HIIT

SUMMARY:
Frailty is defined as a greater susceptibility to stressors resulting from age-related impairments in adaptive biological systems. Frailty leads to poorer physical performance and functional capacity and higher risk of adverse outcomes including falls, hospitalization, and mortality. Resilience, defined as the capacity to recover from disruptions to homeostasis, is critical to successful aging because it precedes frailty and enhances adults' ability to maintain optimal health and function well into older age. Evidence- based therapies to help older adults enhance resilience are limited and the biological underpinnings contributing to improved resilience have not yet been fully characterized. To address this important need, the investigators will conduct a clinical trial to examine the benefits of center- and home-based high intensity interval training (HIIT) on functional capacity, frailty, and resilience, and also to identify novel biomarkers of resilience in older Veterans.

DETAILED DESCRIPTION:
Impact of Home-Based High Intensity Interval Training on Resilience in Older Veterans More than 30% of U.S. Veterans 65 years or older are frail, which is three-times higher than in non-Veterans in the same age group. Frailty is defined as an increased susceptibility to stressors resulting from age-related impairments in adaptive biological systems, leading to higher risk of adverse outcomes including falls, disability, hospitalization, and mortality. Further, frailty prevalence increases with age, affecting 50% of all adults 85 and over. Resilience, which is defined as the capacity to recover from stress-induced disruptions to homeostasis, is critical to successful aging because it precedes frailty and presents an opportunity to intervene on early health deficits, thus preventing aging-related decline in health, function, and quality of life. Evidence-based therapies that enhance resilience in older adults are limited and the complex biological and physiological mechanisms underlying resilience are not yet fully understood. Consequently, Veterans seeking to boost their ability to recover from late-life stressors and prevent frailty have few proven options. The investigators overarching aim is to characterize the complex factors contributing to resilience and develop novel strategies that enhance resilience to boost health span in older adults. Towards this end, the investigators previous VA RR&D SPiRE Award allowed us to demonstrate the feasibility of 12-weeks of high intensity interval training (HIIT) among older Veterans. The investigators successfully enrolled and retained older male and female Veterans and safely conducted individually tailored HIIT that improved cardiorespiratory fitness, lower-body endurance, cognition, and quality of life. The purpose of the proposed larger trial is to build upon the investigators previous successes and develop and implement practical HIIT regimens to reduce frailty and enhance resilience in older Veterans. The investigators will conduct a randomized controlled trial to ascertain the therapeutic benefits of 12-weeks of center- and home-based HIIT on recovery and resilience among Veterans 60 years or older. The investigators have identified a series of biomarkers of resilience and are also seeking to examine key biological drivers of recovery at the molecular level. The investigators proposed study will not only identify feasible methods to measure resilience in older Veterans but will also assess the benefits of home-based HIIT on physical and cognitive performance, frailty, resilience, and health span.

ELIGIBILITY:
Inclusion Criteria:

* Ages 65 years and older
* Male and female, any race
* Medically cleared for exercise
* Non-frail or pre-frail (frailty score < 3)
* Ability to use a recumbent exercise bike

Exclusion Criteria:

* Severe co-morbidity: COPD (GOLD stage IV), CKD ( stage 3)), severe HTN (180 mmHg/120 mmHg)
* VA-SLUMS score 20 or lower (Cognition)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — 157 male and 43 female participants divided equally between non-frail and pre-frail individuals, based upon Fried frailty criteria.
Enrollment: 200 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Sub-maximal oxygen uptake test (VO2max) | Change from baseline to endpoint at 12 weeks
  Participants are asked to exercise on an upright exercise bike as the resistance increases over time. During the exercise, participants are asked to breath through a mask that is connected to a oxygen and carbon dioxide measuring device. The assessment last for approximately 5-10 minutes and provides data the pertain to an individuals lung capacity, breathing rate, and endurance.

SECONDARY OUTCOMES:
Cognitive screen - SLUMS | Change from baseline to endpoint at 12 weeks
  Cognitive status will be assessed using the VA - St. Louis University Mental Survey (VA-SLUMS) involving memory tests, shape recognition, and story recall. The survey scores range from 0-30, with a higher score representing greater cognitive capability. The investigators will also utilize the Cognivue to assess cognition. This is a combinatorial visual and reaction time test.
Amyloid beta 42/40 ratio | Change from baseline to endpoint at 12 weeks
  Serum cognitive marker: change in amyloid beta 42/40 ratio (a unitless measure derived from the ratio of serum amyloid-beta 42 in picograms per milliliter divided by serum amyloid-beta 40 in picograms per milliliter) from baseline to endpoint after 12 weeks.
Cognitive screen - Cognivue | Change from baseline to endpoint at 12 weeks
  Cognivue to assess cognition. This is a computer based combinatorial visual and reaction time test, which is scored 0 to 100.
Phosphorylated tau (P-tau) | Change from baseline to endpoint at 12 weeks
  Serum cognitive marker: plasma levels of phosphorylated tau (P-tau) in picograms per milliliter from baseline to endpoint after 12 weeks.
Brain Derived Neurotrophic Factor (BDNF) | Change from baseline to endpoint at 12 weeks
  Serum cognitive marker: change in Brain Derived Neurotrophic Factor (BDNF) in picograms per milliliter from baseline to endpoint after 12 weeks.
Fatigue | Change from baseline to endpoint at 12 weeks
  Fatigue as assessed by the Brief Fatigue Inventory, which contains 9 self-rated questions with an aggregate score range of 0 to 90.
Sleep quantity and stages | Change from baseline to endpoint at 12 weeks
  Objectively measure sleep quantity and stages using FITBIT Charge 5 actigraphy devices. These devices are worn on the wrist and sleep metrics, including total sleep time and time spent in light, deep, and REM sleep stages.
Sleep quality | Change from baseline to endpoint at 12 weeks
  Sleep quality as assessed by Pittsburgh Sleep Quality Index (PSQI). The PSQI contains 19 self-rated questions that combined to form 7 component scores, each with a range of 0 to 3 points. These in turn are added to yield a global score with a range of 0 to 21 points.
Sleep chronotype | Change from baseline to endpoint at 12 weeks
  Sleep chronotype as assessed by the Morningness/Eveningness survey, which contains 19 self-rated questions with an aggregate score range of 19 to 72.
Sleepiness | Change from baseline to endpoint at 12 weeks
  Sleepiness as assessed by the Epworth Sleepiness Scale, which contains 8 self-rated questions with an aggregate score range of 0 to 24.
Insomnia | Change from baseline to endpoint at 12 weeks
  Insomnia as assessed by the Insomnia Severity Index, which contains 7 self-rated questions with an aggregate score range of 0 to 28.
Anxiety and depression | Change from baseline to endpoint at 12 weeks
  Anxiety and depression as assessed by the Hospital Anxiety and Depression Scale (HADS), which contains 14 self-rated questions with an aggregate score range of 0 to 21.
Sleep disorders | Change from baseline to endpoint at 12 weeks
  Sleep disorders as assessed by the Holland Sleep Disorders Questionnaire, which contains 32 self-rated questions with an aggregate score range of 32 and 160.
30 second chair rise test | Change from baseline to endpoint at 12 weeks
  The investigators will measure endurance in participants by asking participants to sit and rise repeated from a chair as many times in a 30 second time frame.
Frailty assessment | Change from baseline to endpoint at 12 weeks
  Frailty is a syndrome marked by greater susceptibility to adverse outcomes like falls and disability. The investigators will be using the Fried Frailty Phenotype that includes: 1) unexpected weight loss of 5% or more in the last year or BMI < 18.5; score 0 or 1 if positive, 2) grip strength with BMI dependent cut points for men and women; score 0 or 1 if positive, 3) gait speed with height and sex dependent cutoffs; score 0 or 1 if positive, 4) activity assessed by a survey of the frequency of mild/moderate/energetic physical activity; score of 0 or 1, the latter if positive for hardly ever or never engaging in moderate or energetic physical activity, and 5) endurance assessed by survey of bed rest during the day; score of 0 or 1, the latter if occurring every day or every week. The composite score is therefore 0 to 5.
Gait speed | Change from baseline to endpoint at 12 weeks
  Participants are asked to perform a timed walk of approximately 15 feet in length
Arm curl endurance | Change from baseline to endpoint at 12 weeks
  Participants will receive a free weight (8lbs for men and 5lbs for women) and asked to perform total number of arm curls in 30 seconds while in a seated position.
Quality of life assessment | Change from baseline to endpoint at 12 weeks
  Quality of life assessment is performed using the Quality of life, enjoyment, and satisfaction questionnaire - short form (Q-LES-Q-SF) survey instrument. The survey instrument scores from 0 to 70 with a greater score representing better quality of life.
Body Composition (Lean and fat mass) | Change from baseline to endpoint at 12 weeks
  Body composition will be measured using bioelectric impedance (BIA) - a technique where participants are asked to stand on the measurement device and hold on to two metal handles. A light - and non-detectable - current is then transmitted allowing for collection of body fat and lean mass in the subject. The assessment takes roughly 2-3 minutes.
Step counts | Change from baseline to endpoint at 12 weeks
  Objectively measure activity using FITBIT Charge 5 actigraphy devices. These devices are worn on the wrist and capture total steps.
C-Reactive Protein | Change from baseline to endpoint at 12 weeks
  Chronic inflammation may be indicative of distress and lead to chronic diseases. The study will examine the change in C-reactive protein in picograms per milliliter in serum from baseline to endpoint at 12 weeks.
Interleukin-6 | Change from baseline to endpoint at 12 weeks
  Chronic inflammation may be indicative of distress and lead to chronic diseases. The study will examine the change in interleukin-6 in picograms per milliliter in serum from baseline to endpoint at 12 weeks.
Interleukin-10 | Change from baseline to endpoint at 12 weeks
  Chronic inflammation may be indicative of distress and lead to chronic diseases. The study will examine the change in interleukin-10 in picograms per milliliter in serum from baseline to endpoint at 12 weeks.
Eforto Grip endurance | Change from baseline to endpoint at 12 weeks
  participants will be ask to perform a grip endurance assessment using an Eforto device. The device has a squeezable ball that measures force through changes in air pressure in response to squeezing. Participants are asked to attempt three maximal force tests at 5 seconds each, and then asked to maintain maximal grip for as long as they are able to hold.
Biosway balance assessment | Change from baseline to endpoint at 12 weeks
  Participants are measured for microsway (mm/s) while standing on a Biosway balance device. Participants will be asked to hold balance for 45 seconds while standing comfortably, standing with eyes close, standing with a narrow stance, and standing with a narrow stance with eyes closed.
Resilience to Blood occlusion | Change from baseline to endpoint at 12 weeks
  Participants will be asked to wear a blood pressure cuff while a functional near infrared spectroscopy device measures flow flow in the lower arm. The cuff will be applied to restrict blood flow for 2 minutes, and then released to observe blood oxygenation recovery in the lower arm.
Stroop Color and Word Test | Change from baseline to endpoint at 12 weeks
  Participants will be asked to perform the Stroop color and word test. This test features three sections in which the participant will first read words written in black, then part two name the color of blocks, then the final part name the color of the written words.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce R. Troen, MD, Principal Investigator — Kansas City VA Medical Center, Kansas City, MO
Locations (1):
- Kansas City VA Medical Center, Kansas City, MO, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Final data sets will be made available upon specific request and under an authorized Data Use Agreement. This, in addition to the publications being made available via PubMed Central, will enable validation of results by recipients.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After analysis and completion of study along with subsequent publication of results.
Access Criteria: After analysis and completion of study along with subsequent publication of results.